CLINICAL TRIAL: NCT06470997
Title: Specific Biomarkers of Immune-mediated Hepatitis Secondary to Immune Checkpoint
Brief Title: Specific Biomarkers of Immune-mediated Hepatitis Secondary to Immune Checkpoint Inhibitors
Acronym: Pro-CHILI
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL23_0164
Record Dates: First submitted 2024-06-07; First posted 2024-06-24 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Immune-mediated Hepatitis
Keywords: proteomic analysis; blood biomarker; immune-mediated hepatitis secondary to immune checkpoint inhibitors; idiopathic autoimmune hepatitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CHILI : hepatitis induced by immune checkpoint inhibitors: Patient with immunotherapy-induced hepatitis
  Interventions: Biological: Blood sample collection; Procedure: Liver biopsy
- Control group: idiopathic autoimmune hepatitis: Patient with idiopathic autoimmune hepatitis
  Interventions: Biological: Blood sample collection; Procedure: Liver biopsy

INTERVENTIONS:
Biological: Blood sample collection — 6 collections of 5mL blood samples as part of usual care (pre-inclusion visit at Day-7, inclusion visit at Day 0, visit1 at Day 14, visit2 at Day 28, visit3 at Day 90, visit4 at 6 months) and 5 blood sample collections of 5 mL for proteomic analysis in the context of research (inclusion visit at Day 0, visit1 at Day 14, visit2 at Day 28, visit3 at Day 90, visit4 at 6 months)
Procedure: Liver biopsy — 1 liver biopsy performed as part of routine care and 1 additional sample for research: transparietal needle biopsy under ultrasound identification under local anesthesia by a radiologist, 1 to 2 cm per core taken, 2 cores are taken.

SUMMARY:
Identify specific blood biomarkers for hepatitis induced by immune checkpoint inhibitors in comparison to idiopathic autoimmune hepatitis.

DETAILED DESCRIPTION:
Immune checkpoint inhibitors (ICI) have become a pillar of the oncological therapeutic arsenal. Their mechanism of action is based on the restoration of the innate anti-tumor function of T lymphocytes. This mode of action is also the cause of systemic immune-mediated adverse effects. The most common disorders are endocrine, cutaneous and gastrointestinal. The frequency of hepatic toxicities is estimated between 0.7 and 25% depending on the studies, the cancer treated and the ICI combinations used. Currently the description of these hepatitis is brief in the literature and the mechanism of toxicity is not known. Work has already compared histological damage between immune checkpoint inhibitors (CHILI) and autoimmune hepatitis; The investigators find in CHILI a higher ratio of CD8 + /CD4 + lymphocytes. Apart from these clinical, biological or histological descriptions, knowledge is limited. In particular, there are no known predictive factors or prognoses.

The investigators hypothesize that there are mechanistic differences between checkpoint inhibitors induced liver injury and idiopathic autoimmune liver disease. Proteomic analysis is a powerful tool for functional analysis.

ELIGIBILITY:
Inclusion criteria for patients in the CHILI group:

* Patient > 18 years old
* Patient treated with immune checkpoint inhibitors (ICI) alone or in combination
* Patient suffering from Hepatitis secondary to immune checkpoint inhibitors (ICI) grade 3 or 4 Common Terminology Criteria For Adverse Events (CTCAE)*
* Treatment with corticosteroids or Ursodeoxycholic acid (UDCA) not started, or started less than 30 days ago

  * Grade 3 or 4 hepatitis: increase in transaminases and/or alkaline phosphatases ≥ 5 x Upper Limit of Normal (ULN) or total bilirubin ≥ 3

Inclusion criteria for patients in the control group:

* Patient > 18 years old
* Patient suffering from Primary Biliary Cholangitis (PBC)* or Autoimmune Hepatitis (AIH)** or Primary Sclerosing Cholangitis (PSC) ***

Primary Biliary Cholangitis (PBC)* diagnosis :

Association of at least 2 of the following 3 criteria :

* Cholestasis (PAL > 1.5N, Gamma GT > 3N) chronic (> 6 months) without ultrasound abnormality of the bile ducts.
* M2 type anti-mitochondria Ab > 1/40th
* Characteristic histological lesions (non-suppurative destructive cholangitis) or compatible (portal inflammation, granulomas, ductular proliferation, ductopenia, cholestasis).

  ** AIH diagnosis : ALT > 5 N / Ig G > 1.5 - 2 N or anti-smooth muscle ≥ 1/80 / Interface hepatitis of marked intensity The Hepactic Activity Index (HAI) score makes it possible to confirm the diagnosis when all the diagnostic criteria are not met.

  *** PSC diagnosis: presence of chronic cholestasis (alkaline phosphatase > 1.5 N or GGT > 3 N) and typical abnormalities of the bile ducts on cholangio-MRI (Magnetic Resonance Imaging), and in the absence of cause of secondary sclerosing cholangitis
* Treatment with corticosteroids or Ursodeoxycholic acid (UDCA) not initiated, or started less than 30 days ago

Non-inclusion criteria:

* Impossibility of following the patient during the study period
* Liver biopsy not possible
* Other hepatitis diagnoses
* Failure to obtain consent
* Unemancipated minors, people unable to express their consent
* Non-affiliation to a social security or equivalent scheme,
* Persons placed under judicial protection,
* Person participating in another research including a period of exclusion still in progress.
* Pregnant or breastfeeding women
* De novo or old diagnosis (at the time of a flare-up)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CHILI group: patients with hepatitis induced by immune checkpoint inhibitors Control group: patients with idiopathic autoimmune hepatitis
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-07-17 (Actual); Primary Completion 2027-01-18 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Determination of the area under the ROC (Receiver Operation characteristic) curve for hepatitis. | Baseline
  Sensitivity/specialty curve of blood biomarkers identification and expression level by proteomic analysis, specific to immunotherapy-induced hepatitis (CHILI group), versus idiopathic autoimmune hepatitis (control group).

SECONDARY OUTCOMES:
Determination of the area under the ROC (Receiver Operation characteristic) curve for treatment response | Baseline, day 14, day 28, month 3, month 6
  Sensitivity/specialty curve of blood biomarkers identification and expression level by proteomic analysis, specific to response to treatments corticosteroids, UDCA (Ursodeoxycholic acid) established as part of the care).
Responses to treatments | Day 28
  Response to corticosteroid and UDCA (Ursodeoxycholic acid) treatments being defined as a reduction in liver tests of 50%

CONTACTS AND LOCATIONS:
Overall Officials: Lucy MEUNIER, MD, Study Director — University Hospital, Montpellier
Locations (1):
- CHU de Montpellier, Montpellier, France, France

REFERENCES:
- [Background] De Martin E, Michot JM, Rosmorduc O, Guettier C, Samuel D. Liver toxicity as a limiting factor to the increasing use of immune checkpoint inhibitors. JHEP Rep. 2020 Aug 11;2(6):100170. doi: 10.1016/j.jhepr.2020.100170. eCollection 2020 Dec. PMID 33205034
- [Background] Champiat S, Lambotte O, Barreau E, Belkhir R, Berdelou A, Carbonnel F, Cauquil C, Chanson P, Collins M, Durrbach A, Ederhy S, Feuillet S, Francois H, Lazarovici J, Le Pavec J, De Martin E, Mateus C, Michot JM, Samuel D, Soria JC, Robert C, Eggermont A, Marabelle A. Management of immune checkpoint blockade dysimmune toxicities: a collaborative position paper. Ann Oncol. 2016 Apr;27(4):559-74. doi: 10.1093/annonc/mdv623. Epub 2015 Dec 28. PMID 26715621
- [Background] Peeraphatdit TB, Wang J, Odenwald MA, Hu S, Hart J, Charlton MR. Hepatotoxicity From Immune Checkpoint Inhibitors: A Systematic Review and Management Recommendation. Hepatology. 2020 Jul;72(1):315-329. doi: 10.1002/hep.31227. PMID 32167613
- [Background] Haanen J, Obeid M, Spain L, Carbonnel F, Wang Y, Robert C, Lyon AR, Wick W, Kostine M, Peters S, Jordan K, Larkin J; ESMO Guidelines Committee. Electronic address: clinicalguidelines@esmo.org. Management of toxicities from immunotherapy: ESMO Clinical Practice Guideline for diagnosis, treatment and follow-up. Ann Oncol. 2022 Dec;33(12):1217-1238. doi: 10.1016/j.annonc.2022.10.001. Epub 2022 Oct 18. No abstract available. PMID 36270461
- [Background] Zen Y, Yeh MM. Hepatotoxicity of immune checkpoint inhibitors: a histology study of seven cases in comparison with autoimmune hepatitis and idiosyncratic drug-induced liver injury. Mod Pathol. 2018 Jun;31(6):965-973. doi: 10.1038/s41379-018-0013-y. Epub 2018 Feb 5. PMID 29403081
- [Background] Hountondji L, Ferreira De Matos C, Lebosse F, Quantin X, Lesage C, Palassin P, Rivet V, Faure S, Pageaux GP, Assenat E, Alric L, Zahhaf A, Larrey D, Witkowski Durand Viel P, Riviere B, Janick S, Dalle S, Maria ATJ, Comont T, Meunier L. Clinical pattern of checkpoint inhibitor-induced liver injury in a multicentre cohort. JHEP Rep. 2023 Mar 7;5(6):100719. doi: 10.1016/j.jhepr.2023.100719. eCollection 2023 Jun. PMID 37138674
- [Background] Coukos A, Vionnet J, Obeid M, Bouchaab H, Peters S, Latifyan S, Wicky A, Michielin O, Chtioui H, Moradpour D, Fasquelle F, Sempoux C, Fraga M. Systematic comparison with autoimmune liver disease identifies specific histological features of immune checkpoint inhibitor-related adverse events. J Immunother Cancer. 2022 Oct;10(10):e005635. doi: 10.1136/jitc-2022-005635. PMID 36283734
- [Background] Gudd CLC, Au L, Triantafyllou E, Shum B, Liu T, Nathwani R, Kumar N, Mukherjee S, Dhar A, Woollard KJ, Yone Y, Pinato DJ, Thursz MR, Goldin RD, Gore ME, Larkin J, Khamri W, Antoniades CG, Turajlic S, Possamai LA. Activation and transcriptional profile of monocytes and CD8+ T cells are altered in checkpoint inhibitor-related hepatitis. J Hepatol. 2021 Jul;75(1):177-189. doi: 10.1016/j.jhep.2021.02.008. Epub 2021 Feb 22. PMID 33631227
- [Background] Yoshimura K, Tamano Y, Nguyen Canh H, Zihan L, Le Thanh D, Sato Y, Terashima T, Shimoda S, Harada K. A novel pathologic marker, indoleamine 2,3-dioxygenase 1, for the cholangiopathy of immune checkpoint inhibitors-induced immune mediated hepatotoxicity as adverse events and the prediction of additional ursodeoxycholic acid treatment. Med Mol Morphol. 2023 Jun;56(2):106-115. doi: 10.1007/s00795-022-00344-7. Epub 2023 Jan 4. PMID 36599971